CLINICAL TRIAL: NCT05625360
Title: REmotely-delivered Supportive Programs for Improving Surgical Pain Dnd disTrEss (RESPITE)
Brief Title: REmotely-delivered Supportive Programs for Improving Surgical Pain and disTrEss
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB00083414; WFBCCC 98422 (Other: Wake Forest Baptist Comprehensive Cancer Center); R01CA266995 (NIH)
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Pain, Acute; Postoperative Depression; Anxiety; Sleep Disturbance; Malignant Female Reproductive System Neoplasm
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Parasomnias | interventions — Respiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - eHealth Mindful Movement and Breathing Group (eMMB) (Experimental): Participants will be given access to 20-minute eMMB videos (either saved as a local files on an iPad or via links to watch on their own devices) with written instructions for eMMB and to watch a video at least once before surgery (videos have the same content, one is taught in a bed and one in a chair). The instructor will call participants before surgery to offer guidance upon request and meet with participants individually via a synchronous videoconference or telephone session, postoperative day 1 (the day after surgery), or as soon as feasible.
  Interventions: Other: eHealth Mindful Movement and Breathing; Other: PROMIS Questionnaires
- Arm 2 Life Impacts Reflection Group (LIR) (Active Comparator): The format for interactions with an LIR interventionist, frequency of recommended home practice (brief diary entries), and home assessments will be matched to the eMMB group. LIR will not include active ingredients of eMMB.
  Interventions: Other: Life Impacts Reflection; Other: PROMIS Questionnaires

INTERVENTIONS:
Other: eHealth Mindful Movement and Breathing — The self-directed intervention includes an approximately 20-minute eMMB will teach synergistic components: (a) Mindful Meditation - 2 minutes of observing the current state of the body, emotions, thoughts, energy, and breath. Mindful attention may facilitate safe physical movements; (b) Mindful Movement - 10 minutes of gentle movements coordinated with and intended to enhance the breath; (c) Breathing and Relaxation - 3 minutes of placing the hands above the navel (rather than on the belly to avoid discomfort) and noticing them rise and fall with a focus on slightly extending the exhale, which will prepare participants for meditation); (d) Meditation - 5 minutes of observing the natural breath without reacting to it.
  Arms: Arm 1 - eHealth Mindful Movement and Breathing Group (eMMB)
Other: Life Impacts Reflection — This self-directed intervention will focus on active listening, reflection of statements, and avoiding negative judgments. Participants will write brief diary entries daily for four weeks postoperatively and as they choose thereafter. Participants will be given the option of completing diaries on the tablet computer or paper. The instructions for daily diary entries will be, "What were some of the events or circumstances that affected you in the past day? Think back over the past day and write down on the lines below up to five events that had an impact on you." A study team member will call participants to encourage diary completion two days (Postop Day 3) and two weeks after the synchronous session.
  Arms: Arm 2 Life Impacts Reflection Group (LIR)
Other: PROMIS Questionnaires — Various PROMIS questionnaires will be completed by participants (Pain Interference, Sleep Disturbance, Physical Function, Anxiety and Depression)

SUMMARY:
The purpose of this research study is to learn how two different supportive programs may help women feel better after surgery. This study will measure if one type of supportive program is more useful than the other for improving wellbeing after surgery.

DETAILED DESCRIPTION:
Primary Objective: To determine efficacy of eHealth Mindful Movement and Breathing (eMMB) as compared to Life Impact Reflection (LIR) for improving postoperative pain intensity 4-weeks postoperative in patients who received abdominal surgery for a suspected gynecologic malignancy.

Secondary Objectives:

* At week 2 and 3 months post-operative, to determine efficacy of eHealth Mindful Movement and Breathing as compared to LIR for improving pain intensity in patients who received abdominal surgery for a suspected gynecologic malignancy.
* At week 2, week 4, and 3 months postoperative, to determine efficacy of eHealth Mindful Movement and Breathing as compared to LIR for improving affective pain in patients who received abdominal surgery for a suspected gynecologic malignancy.
* To determine efficacy of eHealth Mindful Movement and Breathing as compared to LIR for improving post-operative acute pain (pain intensity within 1 week post-surgery) in patients who received abdominal surgery for a suspected gynecologic malignancy.
* At week 2, week 4, and 3 months postoperative, to determine efficacy of eHealth Mindful Movement and Breathing as compared to LIR for improving pain interference in patients who received abdominal surgery for a suspected gynecologic malignancy.
* At week 2, week 4, and 3 months postoperative, to determine efficacy of eHealth Mindful Movement and Breathing as compared to LIR for improving psychological distress symptoms (i.e., depression) in patients who received abdominal surgery for a suspected gynecologic malignancy.
* At week 2, week 4, and 3 months postoperative, to determine efficacy of eHealth Mindful Movement and Breathing as compared to LIR for improving psychological distress symptoms (i.e., anxiety) in patients who received abdominal surgery for a suspected gynecologic malignancy.
* At week 2, week 4, and 3 months postoperative, to determine efficacy of eHealth Mindful Movement and Breathing as compared to LIR for improving sleep disturbances in patients who received abdominal surgery for a suspected gynecologic malignancy.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form
* Participants age 18 years and older at time of consent.
* Scheduled for an abdominal gynecological surgery (i.e., uterine, ovarian) to remove a mass that is suspected to be malignant
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Able to understand, read and write English (since the intervention is conducted in English)

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Presence of a psychotic disorder, current suicidal ideation, or other unstable major psychiatric condition documented by diagnosis in the medical chart.
* Unwillingness or inability to follow study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Scores - PROMIS Pain Intensity Questionnaire | 4 weeks postoperatively
  Efficacy of the intervention will be evaluated by measuring pain intensity scores between the two groups from the Patient Reported Outcomes Measurement Information System (PROMIS) pain intensity item (How would you rate your pain on average?), which is validated for assessing pain on a numeric rating scale from 0 (no pain) to 10 (worst imaginable pain). Models will be adjusted for the three randomization stratification variables (study site, type of cancer, type of surgery). Linear contrasts will be used to estimate the difference between the two groups.

SECONDARY OUTCOMES:
Change in Pain Intensity - PROMIS Pain Intensity Questionnaire | At 2 weeks and 3 months postoperatively
  Efficacy of the intervention in measuring pain intensity scores from the Patient Reported Outcomes Measurement Information System (PROMIS) pain intensity item (How would you rate your pain on average?), which is validated for assessing pain on a numeric rating scale from 0 (no pain) to 10 (worst imaginable pain). Models will be adjusted for the three randomization stratification variables (study site, type of cancer, type of surgery). Linear contrasts will be used to estimate the difference between the two groups.
Change in Affective Pain - PROMIS Questionnaire | At baseline and 2 weeks, 4 weeks and 3 months postoperatively
  Efficacy of the intervention in affective pain will be assessed with one item (numeric rating scale) on a scale from 0 (not bad at all) to 10 (the most unpleasant feeling possible for me). Models will be adjusted for the three randomization stratification variables (study site, type of cancer, type of surgery). Linear contrasts will be used to estimate the difference between the two groups.
Change in Postoperative Acute Pain - PROMIS Questionnaire | At baseline and 2 weeks, 4 weeks and 3 months postoperatively
  Efficacy of the intervention in post-operative acute pain is defined as pain experienced daily over the first week after surgery and will be measured daily using the PROMIS pain intensity item - (How would you rate your pain on average?), which is validated for assessing pain on a numeric rating scale from 0 (no pain) to 10 (worst imaginable pain). Models will be adjusted for the three randomization stratification variables (study site, type of cancer, type of surgery). Linear contrasts will be used to estimate the difference between the two groups.
Change in Pain Interference | At baseline and 2 weeks, 4 weeks and 3 months postoperatively
  Efficacy of the intervention in improving pain interference will be adjusted for the three randomization stratification variables (study site, type of cancer, type of surgery). Linear contrasts will be used to estimate the difference between the two groups.
Emotional Distress-Depression - Short Form 4a Questionnaire | At baseline and 2 weeks, 4 weeks and 3 months postoperatively
  Efficacy of the intervention in improving psychological distress symptoms will be adjusted for the three randomization stratification variables (study site, type of cancer, type of surgery). Linear contrasts will be used to estimate the difference between the two groups. Scoring scale: 0 - never to 5 - always. The higher the score the greater the depression.
Anxiety- Short Form 4a Questionnaire | At baseline and 2 weeks, 4 weeks and 3 months postoperatively
  Efficacy of the intervention in improving psychological distress symptoms will be adjusted for the three randomization stratification variables (study site, type of cancer, type of surgery). Linear contrasts will be used to estimate the difference between the two groups. Scoring scale: 0 - never to 5 - always. The higher the score the greater the anxiety.
Sleep Disturbance Short Form 4a Questionnaire | At baseline and 2 weeks, 4 weeks and 3 months postoperatively
  Efficacy of the intervention in improving sleep disturbances will be adjusted for the three randomization stratification variables (study site, type of cancer, type of surgery). Linear contrasts will be used to estimate the difference between the two groups. Likert scoring scale: 5 - very poor to 1 - very good or reversed with 5 - not at all to 1 - very much.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J Sohl, PhD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Atrium Health - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No